CLINICAL TRIAL: NCT04475263
Title: Cognitive, Behavioural and Blood Biomarker Assessment After Carbon Monoxide (CO) Exposure
Brief Title: Cognitive and Blood Biomarker Assessment After CO Exposure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St George's, University of London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.0375
Record Dates: First submitted 2020-03-20; First posted 2020-07-17 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carbon monoxide exposure: Confirmed exposure to carbon monoxide

SUMMARY:
Carbon monoxide (CO) is reported to cause around 30 deaths, 200 admissions and 4000 presentations to Emergency Departments each year in the UK. In the longer term, CO poisoning is recognised to cause persistent neurological problems (including impairments of thinking and behavioural changes), which can develop days to weeks after the initial exposure. However, the incidence of these long-term sequelae is unknown. In addition, there is evidence of long-lasting inflammatory changes in the brain and on-going brain cell injury, although how long this persists is also unknown.

Initial assessments of CO exposure can be unreliable if blood tests are not carried out within a relatively short period after the exposure and other biomarkers (such as imaging) are insensitive to detecting previous CO exposure. Certain proteins that are found in brain cells can be detected in the blood of individuals following brain injury and brain cell death. These proteins have been found to be raised in the acute period after minor head injury, persistently raised in patients with a traumatic brain injury and evidence of on going neurodegeneration (i.e. on going brain cell death) and in patients with various types of dementia.

The investigators will assess the presence of these proteins in the blood of 50 participants with proven CO exposure in the sub-acute to chronic timescale (2 weeks to 2 years). This has not been done before and will allow assessment of the presence of on going brain injury in these participants. The investigators will also assess cognitive (e.g. memory, attention and speed of thinking) and behavioural impairments in these participants to help characterise the common impairments suffered following CO exposure and relate these to evidence of persistent brain injury and severity of CO exposure.

ELIGIBILITY:
Inclusion Criteria:

Individuals identified as having confirmed exposure to CO between 2 weeks to 2 years at time of assessment. CO exposure determined by either;

* documented COHb levels above 1.6% in non-smokers and above 6.3% in smokers.
* or, individuals with evidence of being exposed to raised levels of CO and symptoms

Exclusion Criteria:

* age <18 years
* actual or suspected smoke inhalation
* significant neurological or psychiatric illness prior to CO exposure
* inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 individuals with confirmed evidence of CO exposure will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood biomarker level of neurofilament light in participants with proven CO exposure. | 18 months
  Plasma levels of neurofilament light will be measured

SECONDARY OUTCOMES:
Blood biomarker level of tau in participants with proven CO exposure. | 18 months
  Plasma levels of tau will be measured
Blood biomarker level of glial fibrillary acidic protein in participants with proven CO exposure. | 18 months
  Plasma levels of glial fibrillary acidic protein will be measured
Behavioural questionnaire: depression (Patient Health Questionnaire - part 9) | 18 months
  Participants will be asked to complete a validated questionnaire assessing fatigue, depression, anxiety, post-traumatic stress symptoms, problems with attention, quality of life, return to work and illness perceptions. All questionnaires provide a numerical score.
Behavioural questionnaire: anxiety (Generalised Anxiety Disorder Questionnaire - GAD7) | 18 months
  Participants will be asked to complete validated questionnaires assessing fatigue, depression, anxiety, post-traumatic stress symptoms, problems with attention, quality of life, return to work and illness perceptions. All questionnaires provide a numerical score.
Behavioural questionnaire: post-traumatic stress symptoms (Impact of Events Scale) | 18 months
  Participants will be asked to complete validated questionnaires assessing fatigue, depression, anxiety, post-traumatic stress symptoms, problems with attention, quality of life, return to work and illness perceptions. All questionnaires provide a numerical score.
Behavioural questionnaire: Attentional behaviour (Rating Scale of Attentional Behaviour) | 18 months
  Participants will be asked to complete validated questionnaires assessing fatigue, depression, anxiety, post-traumatic stress symptoms, problems with attention, quality of life, return to work and illness perceptions. All questionnaires provide a numerical score.
Behavioural questionnaire: fatigue (Visual Analogue Scale of Fatigue) | 18 months
  Participants will be asked to complete validated questionnaires assessing fatigue, depression, anxiety, post-traumatic stress symptoms, problems with attention, quality of life, return to work and illness perceptions. All questionnaires provide a numerical score.
Behavioural questionnaire: Quality of life (The Short Form (36) Health Survey) | 18 months
  Participants will be asked to complete validated questionnaires assessing fatigue, depression, anxiety, post-traumatic stress symptoms, problems with attention, quality of life, return to work and illness perceptions. All questionnaires provide a numerical score.
Behavioural questionnaire: return to work/social activities (Work and Social Adjustment Scale) | 18 months
  Participants will be asked to complete validated questionnaires assessing fatigue, depression, anxiety, post-traumatic stress symptoms, problems with attention, quality of life, return to work and illness perceptions. All questionnaires provide a numerical score.
Cognitive assessment | 18 months
  Participants will complete a battery of cognitive assessments with a large normative control population. Cognitive tests will assess speed of information processing, reasoning, memory and visuospatial abilities. All results will be a numerical result.

CONTACTS AND LOCATIONS:
Overall Officials: Peter O Jenkins, PhD, Principal Investigator — St. George's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification. Proposals should be directed to peter.jenkins1@nhs.net. To gain access, data requestors will need to sign a data access agreement.
Time Frame: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.
Access Criteria: Researchers who provide a methodologically sound proposal.

DOCUMENTS (1):
  • Study Protocol (2019-12-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT04475263/Prot_000.pdf